CLINICAL TRIAL: NCT01586884
Title: Study to Determine the Safety and Feasibility of Utilizing the CD Leycom Pressure/Conductance Catheter to Determine Optimal LV Pacing Site
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-3-LGH
Record Dates: First submitted 2012-04-20; First posted 2012-04-27 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: LV Pacing; LV Lead Placement; LV Pacing Site; CRT Device Placement
MeSH Terms: conditions — Heart Failure | interventions — Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Ten patients undergoing LV lead placement for either initial CRT device implant or revision of an existing system at Lancaster General Hospital who meet the inclusion and exclusion criteria will be screened and approached for enrollment in this safety and feasibility study. Study participants may have ischemic or non-ischemic cardiomyopathy; results for ischemic and non-ischemic patients will be analyzed separately. Any device system from any manufacturer may be used; the choice of device and leads will be at the implanting physician's discretion.
  Post implant procedures will be the same as those for any CRT implant. Outpatient follow-up other than the 1-month follow-up will be per the implanting physician's usual practice.
  Interventions: Procedure: Pressure/Conductance Catheter

INTERVENTIONS:
Procedure: Pressure/Conductance Catheter — The physician will obtain right femoral arterial access and advance the pressure/conductance catheter to the LV utilizing the retrograde approach. Baseline dP/dt and stroke volume will be recorded in the patient's presenting rhythm.
  The dP/dt and stroke volume will be measured during biventricular pacing. Hemodynamic measurements will be made with the tip of the pacing lead in the distal vessel, followed by repeat measurements with the lead positioned in the mid and proximal portions of the initially selected vein.
  The pacing and hemodynamic measurements will be repeated with the CS lead positioned in two additional veins (if possible). The pressure/conductance catheter will be removed from the left ventricle after 30 minutes, regardless of the number of pacing sites identified/tested. The physician will make the choice of the LV lead placement based on the information gathered up to that point.
  Other Names: CD Leycom Pressure/Conductance Catheter

SUMMARY:
It is hypothesized that it is both safe and feasible to use an interventional approach to LV lead placement (placing the LV lead guided by acute hemodynamic measurements), and that the LV lead can be placed in a position that is superior to the initial empiric lateral wall LV lead location in less than 30 minutes without significant risk to patients. The time from RV capture to LV activation correlates with the optimal pacing site based on stroke volume & dP/dt measurements.

DETAILED DESCRIPTION:
Background

Cardiac synchronization therapy (CRT) is recognized as effective adjunctive therapy for heart failure; however, up to 40% of patients who undergo CRT device placement do not have a favorable response to therapy and are labeled non-responders. The lateral wall of the left ventricle (LV) is generally regarded as the optimal site for LV lead placement and some non-responders with LV leads not on the lateral wall can be converted to responders by repositioning the LV lead to the lateral wall. However, recent studies indicate that in some patients LV lead placement at a site other than the lateral wall may result in a better response to CRT. In such circumstances, empiric lateral wall lead positioning/repositioning may expose patients to the risks of another invasive procedure (including an increased risk of infection); in the case of lead repositioning to improve response to CRT the additional risk is doubled, as there is no certainty that the new position will be superior to the old.

Several investigators have used the acute hemodynamic response to biventricular pacing to determine the optimal LV lead position. To make these measurements some groups used a Millar pigtail catheter (Millar Instruments, Houston, Texas) while other groups used real-time pressure volume loops with a combined pressure-conductance catheter (CD Leycom, Zoetermeer, the Netherlands). One criticism of this method is that acute hemodynamic measurements may not correlate to long term response. However, Delnoy et al demonstrated that acute improvements in LV function as measured by pressure-volume loops during implantation corresponded to clinical and echocardiographic improvement during follow-up. In addition, Duckett et al demonstrated that the acute dP/dt response to LV pacing is useful for predicting which patients are likely to remodel in response to CRT, for both dilated and ischemic cardiomyopathy.

Despite these observations, few practitioners routinely utilize acute hemodynamic measurements for LV lead placement at the time of device implantation. Many practitioners believe targeted LV lead placement is impractical due to the time required to determine hemodynamic response to CRT and reposition the LV lead, and that venous anatomy, phrenic nerve pacing, and high pacing thresholds severely limit options for LV lead placement.

Study Hypothesis

It is hypothesized that it is both safe and feasible to use an interventional approach to LV lead placement (placing the LV lead guided by acute hemodynamic measurements), and that the LV lead can be placed in a position that is superior to the initial empiric lateral wall LV lead location in less than 30 minutes without significant risk to patients. The time from RV capture to LV activation correlates with the optimal pacing site based on stroke volume & dP/dt measurements.

Study Purpose

The purpose of this study is to determine whether utilizing the CD Leycom pressure-conductance catheter to measure dP/dt and pressure volume loops at the time of LV lead implant (whether for the initial CRT implant or revision of an existing system) is both safe and feasible. It is hoped that the study will determine whether it is possible to use a patient's hemodynamic response to pacing to locate an LV pacing site that provides better hemodynamic response to CRT than the empirically selected lateral wall pacing site without significant patient risk (in terms of radiation exposure, amount of contrast received, procedure time, potential injury).

ELIGIBILITY:
Inclusion Criteria

1. Ischemic or non-ischemic cardiomyopathy
2. Patient meets all current criteria for CRT (NYHA Class III-IV heart failure, QRS ≥ 120 ms, LVEF ≤ 35%, optimal medical therapy).
3. Patient willing/able to sign study informed consent and HIPAA authorization.

Exclusion Criteria

1. Patient does not meet current criteria for CRT implant
2. Mechanical aortic valve
3. Left ventricular thrombus
4. Aortic stenosis
5. No palpable femoral pulse
6. Extensive atherosclerotic disease of the aorta
7. Serum creatinine > 2.5
8. Patient not willing/able to sign study informed consent/HIPAA authorization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Feasibility | 30 Minutes
  Feasibility of measuring dP/dt in a maximum of 3 veins within 30 minutes.
Procedure time | 2 Hours
  Additional procedure time for pressure measures.
Radiation exposure | 2 Hours
  During procedure as measured with Gafchromic film.
Contrast nephropathy | 2 Hours
  From procedure.
Death | 1 Month
  From procedure.

SECONDARY OUTCOMES:
Feasibility | 1 Month
  The secondary endpoint for the study is to determine the percentage of patients in whom the empirically selected "best" lateral wall LV lead location was the best site based on the hemodynamic measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Worley, MD, Study Chair — Lancaster General Hospital; Susan A Deck, BS RN, Principal Investigator — Lancaster General Hospital; Douglas Gohn, MD, Principal Investigator — Lancaster General Hospital; Kay M Knepper, RN, Principal Investigator — Lancaster General Hospital; Kruse Lou Anne, RN, Principal Investigator — Lancaster General Hospital; McKernan Pulliam Melissa, MD, Principal Investigator — Lancaster General Hospital; Pulliam Ward, MD, Principal Investigator — Lancaster General Hospital; Testa Heidi, RN, Principal Investigator — Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Spragg DD, Dong J, Fetics BJ, Helm R, Marine JE, Cheng A, Henrikson CA, Kass DA, Berger RD. Optimal left ventricular endocardial pacing sites for cardiac resynchronization therapy in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2010 Aug 31;56(10):774-81. doi: 10.1016/j.jacc.2010.06.014. PMID 20797490
- [Background] Derval N, Steendijk P, Gula LJ, Deplagne A, Laborderie J, Sacher F, Knecht S, Wright M, Nault I, Ploux S, Ritter P, Bordachar P, Lafitte S, Reant P, Klein GJ, Narayan SM, Garrigue S, Hocini M, Haissaguerre M, Clementy J, Jais P. Optimizing hemodynamics in heart failure patients by systematic screening of left ventricular pacing sites: the lateral left ventricular wall and the coronary sinus are rarely the best sites. J Am Coll Cardiol. 2010 Feb 9;55(6):566-75. doi: 10.1016/j.jacc.2009.08.045. Epub 2009 Nov 20. PMID 19931364
- [Background] Delnoy PP, Ottervanger JP, Vos DH, Elvan A, Misier AR, Beukema WP, Steendijk P, van Hemel NM. Upgrading to biventricular pacing guided by pressure-volume loop analysis during implantation. J Cardiovasc Electrophysiol. 2011 Jun;22(6):677-83. doi: 10.1111/j.1540-8167.2010.01968.x. Epub 2010 Dec 6. PMID 21134027
- [Background] Duckett SG, Ginks M, Shetty AK, Bostock J, Gill JS, Hamid S, Kapetanakis S, Cunliffe E, Razavi R, Carr-White G, Rinaldi CA. Invasive acute hemodynamic response to guide left ventricular lead implantation predicts chronic remodeling in patients undergoing cardiac resynchronization therapy. J Am Coll Cardiol. 2011 Sep 6;58(11):1128-36. doi: 10.1016/j.jacc.2011.04.042. PMID 21884950